CLINICAL TRIAL: NCT05803434
Title: Open-label Pilot Study to Assess the Efficacy and Safety of Cannabidiol Oral Solution as an Adjunctive Treatment for Children and Young Adults With Rare Disease-associated Severe Epilepsy
Brief Title: Cannabidiol in Children and Young Adults With Rare Disease-associated Severe Epilepsy
Acronym: CBD_RE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Renzo Guerrini, Director, Head of Child Neurology Department, Principal Investigator, Clinical Professor, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBD_RE
Record Dates: First submitted 2023-02-28; First posted 2023-04-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Epilepsy; Rare Diseases
Keywords: drug resistant epilepsy; rare epilepsy; cannabidiol
MeSH Terms: conditions — Epilepsy; Rare Diseases; Drug Resistant Epilepsy | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cannabidiol treatment (Experimental)
  Interventions: Drug: Cannabidiol oral solution

INTERVENTIONS:
Drug: Cannabidiol oral solution — Cannabidiol will be administered orally twice daily into equally divided doses. The starting dose is 2.5 mg/kg twice daily. The dose can be gradually increased to 5 mg/kg twice daily, which is the recommended maintenance dose, up to a maximum dose of 10 mg/kg twice daily, according to tolerability and clinical response.
  Following titration, subjects will continue treatment over a 20-week maintenance period. The total treatment duration from the beginning of the titration period till the end of the maintenance period will be 24 weeks.

SUMMARY:
This is a pilot, open-label, phase II study. The main objective of the study is to demonstrate that Cannabidiol (CBD), used in addition to current anti-seizure medications (ASMs) reduces the number and/or severity of motor (generalized, focal, or both) seizures in children and young adults with rare disease-associated severe epilepsy.

Secondary objectives include assessment of safety and tolerability, changes in behaviour, cognition and sleep, pharmacokinetic interaction with concurrent ASMs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female;
2. Children (age 2-18 years) and young adults (18-25 years), as of the day of the Screening Visit;
3. Subject with rare disease-associated severe epilepsy. Subject has been certified by the National Health System as affected by a rare disease listed in https://www.malattierare.gov.it
4. Patient has severe epilepsy, with at least 4 motor (generalized, focal, or both) seizures per month during baseline period, despite 2 or more current or prior ASMs;
5. Previous treatment with at least 2 ASMs;
6. Currently taking at least 1 other ASMs or between one and four ASMs, with a stable antiseizure treatment for the previous 4 weeks (including ketogenic diet and vagal nerve stimulation);
7. Subject's parent/caregiver has been informed of the nature of the study and informed consent has been obtained from the legally responsible parent/guardian;
8. Subject's parent/caregiver is willing and able to be compliant with diary completion, visit schedule and study drug accountability in the opinion of the investigator

Exclusion Criteria:

1. Age <2 years;
2. Known hypersensitivity to CBD or any of the excipients in the study formulation;
3. Progressive neurological disease;
4. Clinically significant unstable medical conditions other than epilepsy that may place patient's safety at risk;
5. Any other significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, may influence the result of the study, or affect the patient's ability to participate in the study;
6. Impaired hepatic function at screening defined as any of the following: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3 times the upper limit of normal (ULN) and total bilirubin (TBL) greater than 2 times the ULN;
7. Subject taking more than four concurrent ASMs;
8. Subject has taken corticotropins in the six months prior to screening;
9. Subjects taking felbamate, and they have been taking it for less than one year prior to screening;
10. Inadequate supervision by parents and/or caregivers as judged by the investigator;
11. Subject has been part of a clinical trial involving another investigational medicinal product in the previous six months;
12. Current or past use of recreational or medicinal cannabis, or cannabinoid-based medications, within the three months prior to screening and is unwilling to abstain for the duration for the study;
13. Female patients who are pregnant;
14. Female patients of childbearing potential or male patient whose partner is of childbearing potential, unless willing to ensure that they or their partner use a highly effective method of birth control during the study and for three months thereafter.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of generalized and/or focal motor-onset seizure frequency | 24 weeks
  percentage change per 28 days from the 4-week baseline period in generalized and/or focal motor-onset seizure frequency during the 24-week treatment period
Change in severity of generalized and/or focal motor-onset seizure frequency | 24 weeks
  a score will be established for each patient, based on review and comparison of all baseline-EEG/7-weeks control-EEG and baseline-EEG/15-weeks control-EEG, with values ranging from 0 (= worsened EEG), to a maximum of 2 (= improved); 1 will be assigned if the EEG trace is unmodified

SECONDARY OUTCOMES:
Incidence of adverse events | 24 weeks
  Adverse events reporting according to Common Terminology Criteria for Adverse Events (CTCAE) from 1 (mild) to 5 (death)
Body weight | 24 weeks
  Measurement of body weight for tolerability monitoring
Maximum Plasma Concentraion [Cmax] of concurrent ASMs | 24 weeks
  blood levels of concurrent ASMs will be taken at baseline and every 4 weeks
Number of subjects considered treatment responders | 24 weeks
  Number of subjects with a ≥25%, ≥50% ≥75% reduction in motor (generalized, focal, or both) seizures from baseline
Number of subjects who are free of motor (generalized, focal, or both) seizures | 24 weeks
  Number of subjects who are free of motor (generalized, focal, or both) seizures
Longest period of seizure freedom | 24 weeks
  Longest period of seizure freedom
Number of patients experiencing a >25% worsening, -25 to +25% no change, 25-50% improvement, 50-75% improvement or >75% improvement in total seizures from baseline | 24 weeks
  Number of patients experiencing a >25% worsening, -25 to +25% no change, 25-50% improvement, 50-75% improvement or >75% improvement in total seizures from baseline
Changes from baseline in number of inpatient hospitalizations due to epilepsy | 24 weeks
  Changes from baseline in number of inpatient hospitalizations due to epilepsy
Change in severity of seizures will be assessed using a pediatric adaptation of the Chalfont Seizure Severity Scale | 24 weeks
  Change in severity of seizures will be assessed using a pediatric adaptation of the Chalfont Seizure Severity Scale (from 1 minimum severity to >100 max severity)
Change from baseline to 6-months after treatment initiation in number of seizure-free days | 24 weeks
  Change from baseline to 6-months after treatment initiation in number of seizure-free days